CLINICAL TRIAL: NCT02739607
Title: Internet-delivered Transdiagnostic Intervention for Anxiety and Depression in Romania- A Randomized Control Trial
Brief Title: Internet-delivered Transdiagnostic Intervention for Anxiety and Depression
Acronym: iTAD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: West University of Timisoara (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WUTimisoara-iTAD
Record Dates: First submitted 2016-04-12; First posted 2016-04-15 (Estimated); Last update posted 2016-05-06 (Estimated); Status verified 2016-05

CONDITIONS: Depression; Dysthymic Disorder; Panic Disorder; Social Phobia; Specific Phobia; Obsessive-Compulsive Disorder; Generalized Anxiety Disorder
Keywords: emotional disorders; internet-delivered intervention; anxiety; depression; transdiagnostic
MeSH Terms: conditions — Depression; Dysthymic Disorder; Panic Disorder; Phobia, Social; Phobia, Specific; Obsessive-Compulsive Disorder; Generalized Anxiety Disorder; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Transdiagnostic program (Experimental): This arm represents the Transdiagnostic intervention program for emotional disorders. The intervention, based on the Cognitive Behavioral Therapy (CBT) principles, is designed to encourage participants to confront and experience uncomfortable emotions, and use adaptive coping mechanisms.
  Interventions: Behavioral: Transdiagnostic program
- Wait list control group (No Intervention): This arm represents the wait-list comparison group.

INTERVENTIONS:
Behavioral: Transdiagnostic program — This transdiagnostic program is based on the general Cognitive Behavioral Therapy (CBT) principles and targets core higher order factors such as negative affectivity and emotion dysregulation, using common intervention techniques applicable across disorders. The program was designed to directly address the aversive emotional experiences often reported by clients, hoping to reverse participants' maladaptive thinking style and dysfunctional behaviors.
  Arms: Transdiagnostic program

SUMMARY:
Objectives

1. To test the effectiveness and acceptability of an augmented internet-supported transdiagnostic intervention in Romania.
2. To assess the cost-effectiveness of the Internet version of the transdiagnostic program as compared to a standard treatment/usual care.

DETAILED DESCRIPTION:
The effectiveness of a transdiagnostic intervention will be compared with a wait list control group using a randomized control trial (RCT) design in a culture where this has not been tested before. The treatment approach is mainly emotion-focus, teaching participants how to confront and experience uncomfortable emotions, and how more adaptive coping mechanisms could be used. Because internet-delivered interventions represent an effective way to disseminate evidence-based programs, investigators decided to present our intervention online.

ELIGIBILITY:
Inclusion Criteria:

* be fluent in Romanian
* be over 18 years
* have the principal diagnostic of generalized anxiety disorder and/or obsessive-compulsive disorder and/or panic disorder and/or social anxiety disorder and/or major depression disorder and/or dysthymia (or any combination of these diagnostics) on Structured Clinical Interview for the Diagnostic and Statistical Manual for Mental Disorders (SCID-I)
* have access to an Internet connected computer

Exclusion Criteria:

* suicidal ideation
* ongoing psychological treatment for generalized anxiety disorder and/or obsessive-compulsive disorder and/or panic disorder and/or social anxiety disorder and/or major depression disorder and/or dysthymia
* other primary disorder that need treatment
* obstacle to participation (i.e., long travel plans)
* recent change in psychiatric medication (i.e., during the last 6 weeks)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-04; Primary Completion 2016-09 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Penn State Worry Questionnaire (PSWQ) | Absolute values (average score) of PSWQ at 11 weeks (post-intervention)
  The PSWQ was designed to measure participant's level of generalized anxiety or worry. The scale is unidimensional and the total score rages from 16 to 80. Low scores are associated with low levels of worry, while high scores are associated with high levels of worry.
Social Phobia Inventory (SPIN) | Absolute values (average score) of SPIN at 11 weeks (post-intervention)
  The SPIN was designed to measure participant's level of social phobia. The scale is unidimensional and the total score rages from 0 to 68. Low scores are associated with low levels of social phobia, while high scores are associated with high levels of social phobia.
Yale-Brown Obsessive Compulsive Scale (YBOCS) | Absolute values (average score) of YBOCS at 11 weeks (post-intervention)
  The YBOCS was designed to measure participant's level of obsessions and compulsions (O&C). The scale total score rages from 0 to 40. Low scores are associated with low levels of O&C, while high scores are associated with high levels of O&C.
Panic Disorder Severity Scale - Self Report (PDSS-SR) | Absolute values (average score) of PDSS-SR at 11 weeks (post-intervention)
  The PDSS-SR was designed to measure participant's level of panic. The scale is unidimensional and the total score rages from 0 to 28. Low scores are associated with low levels of panic, while high scores are associated with high levels of panic.
Post-Traumatic Stress Disorder Checklist for the Diagnostic and Statistical Manual-5 (PCL-5) | Absolute values (average score) of PCL-5 at 11 weeks (post-intervention)
  The PCL-5 was designed to measure participant's level of post-traumatic stress. The scale is unidimensional and the total score rages from 0 to 80. Low scores are associated with low levels of post-traumatic stress, while high scores are associated with high levels of post-traumatic stress.
Beck Depression Inventory-II (BDI-II) | Absolute values (average score) of BDI-II at 11 weeks (post-intervention)
  The Beck Depression Inventory-II (BDI-II) was designed to measure participant's level of depression. The scale is unidimensional and the total score rages from 0 to 63. Low scores are associated with low levels of depression, while high scores are associated with high levels of depression.

SECONDARY OUTCOMES:
Emotion Regulation Questionnaire (ERQ) | Absolute values (average score) of ERQ at 11 weeks (post-intervention)
  The ERQ was designed to measure participant's level of emotion regulation. The scale is multidimensional and measures two emotion regulation strategies: reappraisal and suppression. Low scores are associated with low levels of emotion regulation, while high scores are associated with high levels of emotion regulation.
Anxiety Sensitivity Index (ASI) | Absolute values (average score) of ASI at 11 weeks (post-intervention)
  The ASI was designed to measure participant's level of anxiety sensitivity. The scale is unidimensional and the total score rages from 0 to 64. Low scores are associated with low levels of anxiety sensitivity, while high scores are associated with high levels of anxiety sensitivity.
Beck Anxiety Inventory (BAI) | Absolute values (average score) of Treatment satisfaction and acceptability at 11 weeks (post-intervention)
  The BAI was designed to measure participant's level of anxiety. The scale is unidimensional and the total score rages from 0 to 63. Low scores are associated with low levels of anxiety, while high scores are associated with high levels of anxiety.
Almost Perfect Scale-Revised (APS-R) | Absolute values (average score) of APS-R at 11 weeks (post-intervention)
  The APS-R was designed to measure participant's level of perfectionism. The scale is multidimensional and measures three dimensions of perfectionism: high standards, order and discrepancy. Low scores are associated with low levels of perfectionism, while high scores are associated with high levels of perfectionism.

CONTACTS AND LOCATIONS:
Overall Officials: Bogdan T Tulbure, PhD, Study Director — West University of Timisoara
Locations (1):
- West University of Timisoara, Timișoara, Timiș County, Romania

IPD SHARING:
Plan to Share IPD: No
Data will be process only at the group level. No individual data will be shared to third parties.

REFERENCES:
- [Derived] Tulbure BT, Rusu A, Sava FA, Salagean N, Farchione TJ. A Web-Based Transdiagnostic Intervention for Affective and Mood Disorders: Randomized Controlled Trial. JMIR Ment Health. 2018 May 24;5(2):e36. doi: 10.2196/mental.8901. PMID 29798831
- See also: Project official website — http://e-cbt.ro/program/psitad